CLINICAL TRIAL: NCT06962371
Title: GUARDIAN Australian Feasibility Study: Safety and Feasibility
Brief Title: Clinical Feasibility and Evaluation Study of POINT-GUARD Embolic Protection Device During TAVR (GUARDIAN)
Acronym: GUARDIAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Transverse Medical, Inc. (Industry)
Collaborators: Medical Metrics Diagnostics, Inc (Industry); Monash Health (Other); Transverse Medical Australia (Unknown); Ascend Clinical (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CA-0007
Record Dates: First submitted 2025-04-03; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Transcatheter Aortic Valve Implantation (TAVI); Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement
Keywords: CEP; Cerebral Embolic Protection; CEP Device; TAVR; TAVI; stroke
MeSH Terms: conditions — Aortic Valve Stenosis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Point-Guard (Experimental)
  Interventions: Device: cerebral embolic protection

INTERVENTIONS:
Device: cerebral embolic protection — Use of Transverse Medical Inc. Point-Guard CEP device.

SUMMARY:
The purpose of this study is to assess the feasibility and safety of the Transverse Medical, Inc. Point-Guard device. This feasibility study is a limited clinical investigation of the Point-Guard device. The study will be conducted to evaluate the device design concept with respect to clinical safety and device functionality.

DETAILED DESCRIPTION:
This is a prospective, single-arm, multi-center, open study to assess the clinical performance and safety of the Point-Guard CEPD during a TAVR procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is ≥18 years of age;
2. The patient meets indications for Transcatheter Aortic Valve Replacement (TAVR);
3. The patient is willing to comply with protocol-specified follow-up evaluations;
4. The patient has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent, approved by the appropriate Institutional Review Board or Ethics Committee.

Exclusion Criteria:

1. TAVR conducted via other than transfemoral access (subclavian, axillar, transapical, transaortic, carotid or transcaval).
2. Anatomy that precludes safe delivery and retrieval of the investigational device.
3. Current or planned treatment with any investigational drug or investigational device during the study enrollment or follow-up period.
4. Cardiovascular surgical or interventional procedure 10 days prior or planned during the TAVR procedure or during the 30-day study follow-up.
5. Patients with uncontrolled bleeding disorders.
6. Patients who are pregnant, as confirmed by a positive pregnancy test.

General Exclusion Criteria

1. TAVR conducted via other than transfemoral access (subclavian, axillar, transapical, transaortic, carotid or transcaval).
2. Anatomy that precludes safe delivery and retrieval of the investigational device.
3. Current or planned treatment with any investigational drug or investigational device during the study enrollment or follow-up period.
4. Cardiovascular surgical or interventional procedure 10 days prior or planned during the TAVR procedure or during the 30-day study follow-up.
5. Patients with uncontrolled bleeding disorders.

5. Patients who are pregnant, as confirmed by a positive pregnancy test.

Magnetic resonance imaging exclusion criteria:

1. Body Mass Index (BMI) and/or total body weight precluding imaging in scanner.
2. Contraindications to MRI (subjects with any implantable temporary or permanent pacemaker or defibrillator, metal implants in field of view, metallic fragments, clips, or devices in the brain or eye before TAVR procedure).
3. High risk of complete AV block after TAVR, with the need of permanent pacemaker (e.g., subjects with pre-existing bifascicular block or complete right bundle branch block plus any degree of AV block).
4. Existing or planned implantation of a pacemaker or defibrillator implantation within the first 3 days after TAVR.
5. Claustrophobia precluding MRI scanning.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | From beginning of TAVI procedure to end.
  Technical success, defined as successful deployment, positioning and retrieval per the Instructions For Use (IFU), with minimal device interference, and as outlined below:
  * Deployment of the Point-Guard filter unit from the Delivery sheath into the aortic arch;
  * Positioning of the Point-Guard device within the aortic arch;
  * Retrieving and removing the Point-Guard device intact;
  * Minimal device interference (operator assessed).
Primary Safety Endpoints | Beginning of TAVI procedure to 30 days post-procedure.
  1. Primary Safety Endpoint: TAVR procedure complications associated with the delivery, positioning, and removal of the test device.
  2. Primary Safety Endpoint: MACCE (all death, all stroke, and acute kidney injury class 3) within 72 hours or discharge, whatever occurs first and at 30 days.

OTHER OUTCOMES:
Observational Endpoints | 24 hours pre-procedure to 24 hours post-procedure
  1. Reduction in Median Total New Lesion Volume in whole-brain as assessed by traditional 1.5T DW-MRI as soon as possible and within twenty-four (24) hours post-procedure. [Time Frame: Day 0-1 days Post-Procedure]
  - Total new lesion volume is defined as the sum of all diffusion- positive new cerebral lesions in post-TAVR DW-MRI relative to the pre-TAVR DW-MRI scans. (in mm^3)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Gooley, MD, Principal Investigator — Monash Health
Locations (1):
- Victorian Heart Hospital, Clayton, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
IPD to be used for internal device design validation only.